CLINICAL TRIAL: NCT04391179
Title: Dipyridamole to Prevent Coronavirus Exacerbation of Respiratory Status (DICER) in COVID-19
Acronym: DICER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jason Scott Knight, Associate Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00179783
Record Dates: First submitted 2020-05-15; First posted 2020-05-18 (Actual); Results first posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: COVID; Corona Virus Infection; Covid-19; SARS-CoV-2 Infection
Keywords: Oxygen
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dipyridamole 100 Milligram(mg) (Experimental): 100 milligrams (mg) by mouth (PO) four times a day (QID)
  Interventions: Drug: Dipyridamole 100 Milligram(mg)
- Placebo (Placebo Comparator): Placebo given by mouth four times a day
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Dipyridamole 100 Milligram(mg) — Drug will be given for 14 days while in the hospital.
  Arms: Dipyridamole 100 Milligram(mg)
Drug: Placebo oral tablet — Placebo will be given for 14 days while in the hospital.
  Arms: Placebo

SUMMARY:
The most severe manifestations of COVID-19 include respiratory failure, coagulation problems, and death. Inflammation and blood clotting are believed to play an important role in these manifestations. Research in humans has shown that dipyridamole can reduce blood clotting. This research study is being conducted to learn whether 14 days of treatment with dipyridamole will reduce excessive blood clotting in COVID-19.

This study will enroll participants with confirmed coronavirus (SARS-CoV)-2 infection that are admitted. Eligible participants will be randomized to receive dipyridamole or placebo for 14 days in the hospital. In addition, data will be collected from the medical record, and there will also be blood draws during the hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent prior to performing study procedures unless they have a legally authorized representative (LAR)
* Confirmed coronavirus (SARS-CoV-2) infection
* Currently hospitalized or anticipated hospitalization requiring supplemental oxygen

Exclusion Criteria:

* In the opinion of at least two investigators, unlikely to survive for >48 hours from screening
* Concurrent enrollment in a clinical trial with a cytokine inhibitor (targeting interleukin-6 (IL-6), Interleukin-6 Receptor (IL-6R), IL-1, or Janus kinase). Use of remdesivir is permitted.
* Currently on invasive mechanical ventilation.
* Hypotension defined as systolic blood pressure < 90 mmHg on two sequential readings at least 4 hours apart
* Pregnant or breastfeeding
* Concurrent dual antithrombotic therapy (aspirin or P2Y12 inhibitor plus anticoagulation to treat deep venous thrombosis or pulmonary embolism (single antiplatelet or anticoagulant agent at prophylaxis or therapeutic dose is permitted)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) greater than 5 times upper limit of normal, hemoglobin < 8 grams per deciliter (g/dL), or platelets <50,000 per cubic millimeter (mm3)
* History of recent major bleeding, defined in accordance with the criteria of the International Society on Thrombosis and Hemostasis (ISTH).
* Any physical examination findings and/or history of any illness that, in the opinion of the study investigator, might confound the results of the study or pose an additional risk to the patient by their participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2020-05-31 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2021-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Knight, MD, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fischer AL, Messer S, Riera R, Martimbianco ALC, Stegemann M, Estcourt LJ, Weibel S, Monsef I, Andreas M, Pacheco RL, Skoetz N. Antiplatelet agents for the treatment of adults with COVID-19. Cochrane Database Syst Rev. 2023 Jul 25;7(7):CD015078. doi: 10.1002/14651858.CD015078. PMID 37489818

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between May 2020 and January 2021, 99 eligible participants received at least one dose of study drug and were included in the analysis.
Period: Overall Study
Arm/Group | Dipyridamole 100 Milligram(mg) | Placebo
Started | 49 | 50
Completed | 34 | 34
Not Completed | 15 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dipyridamole 100 Milligram(mg) | Placebo | Total
Number analyzed (Participants) | 49 | 50 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 29 | 60
  >=65 years | 18 | 21 | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 33
  Male | 33 | 33 | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 46 | 48 | 94
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 45 | 42 | 87
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
D-Dimer [Mean (Standard Deviation); unit: mg/L] — Baseline plasma D-dimer level Population: Three patients did not have baseline D-Dimer values on the day of study drug.
  mg/L
    number analyzed (Participants) | 47 | 49 | 96
    (all) | 1.06 (.80) | 1.24 (1.46) | 1.15 (1.18)
Oxygen Saturation (SpO2)/Fraction of Inspired Oxygen (FiO2) [Mean (Standard Deviation); unit: ratio] | 308 (70) | 310 (72) | 309 (71)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in D-dimer
Description: average percent daily change in plasma D-dimer levels compared to baseline
Time Frame: baseline, up to approximately 14 days after last study drug administration
Measure: Mean (97.8% Confidence Interval); unit: percent daily change
Arm/Group | Dipyridamole 100 Milligram(mg) | Placebo
Number analyzed (Participants) | 49 | 50
percent daily change | -5.6 [-10.2 to -0.07] | -2.4 [-6.9 to 2.3]
Statistical Analysis 1: Comparison: Dipyridamole 100 Milligram(mg) vs Placebo; Test type: Superiority; p = 0.24, Mixed Models Analysis; Slope = -.033, 95% CI 2-sided [-.089 to .023], Standard Error of Mean .027 — Estimation represents log-scale difference between average daily change in D-Dimer for Dipyridamole patients minus placebo average daily change. Negative estimates indicate that D-Dimer levels decline faster in Dipyridamole versus placebo patients

2. Primary Outcome: Number of Participants With Wins at Each Level of a Hierarchical Composite Rank Score
Description: Compare each dipyridamole patient head to head against each placebo patient using a hierarchical composite rank score
  1. death
  2. days on mechanical ventilation
  3. dichotomized (yes/no) decrease in daily average SpO2/FiO2 of at least 50 units relative to day 1 at anytime during the observation period
  4. cumulative sum of COVID ordinal score during study hospitalization. Ordinal scores could range 1-8. Levels 1 and 2 imply no hospitalization and 8 is the worst possible score (death); by definition, the subjects in the DICER study were hospitalized during the time period in which the study observed their ordinal scores.
Time Frame: up to approximately 30 days after hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Dipyridamole 100 Milligram(mg) | Placebo
Number analyzed (Participants) | 49 | 50
Participants
  Composite endpoint- death | 0 | 3
  Composite endpoint- mechanical ventilation during hospitalization | 3 | 4
  Composite endpoint- 50+ unit drop SpO2/FiO2 | 13 | 11
  Composite endpoint- remaining (ties among patients evaluated by ordinal score) | 33 | 32
Statistical Analysis 1: Comparison: Dipyridamole 100 Milligram(mg) vs Placebo; A win ratio analysis of the hierarchical composite outcome requiring direct comparison of outcomes between each dipyridamole patient and placebo patient. The patient with the superior outcome is adjudicated the 'winner' and receives a +1 score, while the 'loser' scores -1; Test type: Superiority; p = .98, Mantel Haenszel; win ratio = 1.00, 97.8% CI 2-sided [0.78 to 1.29] — win ratio= (the probability of a win for the dipyridamole patient)/(probability of a win for the placebo patient)

3. Secondary Outcome: Days Alive and Free of Organ Support
Description: Organ support is defined as receipt of invasive mechanical ventilation, vasopressor therapy, ECMO support, or dialysis.
Time Frame: up to approximately 28 days after last study drug administration score
Population: 5 participants on dipyridamole and 2 participants on placebo were excluded from this analysis because of their early withdrawal from the study (prior to 28 days after last study drug administration).
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Dipyridamole 100 Milligram(mg) | Placebo
Number analyzed (Participants) | 44 | 48
days | 28 [28 to 28] | 28 [28 to 28]
Statistical Analysis 1: Comparison: Dipyridamole 100 Milligram(mg) vs Placebo; Test type: Superiority; p = .08, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Individual Component of Composite Endpoint- Death
Description: Death of any cause during duration of study participation
Time Frame: up to approximately 30 days after hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Dipyridamole 100 Milligram(mg) | Placebo
Number analyzed (Participants) | 49 | 50
Participants | 0 | 3
Statistical Analysis 1: Comparison: Dipyridamole 100 Milligram(mg) vs Placebo; Test type: Superiority; p = .09, Log Rank

5. Secondary Outcome: Individual Component of Composite Endpoint- Days on Mechanical Ventilation
Description: The number of days spent on invasive mechanical ventilation during study hospitalization.
Time Frame: up to 14 days after study drug administration
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Dipyridamole 100 Milligram(mg) | Placebo
Number analyzed (Participants) | 49 | 50
days | 0.33 (1.36) | 0.88 (2.74)
Statistical Analysis 1: Comparison: Dipyridamole 100 Milligram(mg) vs Placebo; Test type: Superiority; p = 0.36, regression, negative binomial; Mean Difference (Net) = 0.29, 95% CI 2-sided [0.02 to 3.94] — estimated ratio of days on mechanical ventilation for dipyridamole and placebo

6. Secondary Outcome: Individual Component of Composite Endpoint- Sp02/Fi02 (as Shown by Participant Count)
Description: Binary outcome indicating patients whose Sp02/Fi02 dropped 50 points relative to baseline at any time during hospitalization.
Time Frame: up to 14 days after study drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | Dipyridamole 100 Milligram(mg) | Placebo
Number analyzed (Participants) | 49 | 50
Participants | 14 | 14
Statistical Analysis 1: Comparison: Dipyridamole 100 Milligram(mg) vs Placebo; Test type: Superiority; p = .94, Regression, Logistic; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.43 to 2.51] — Odds of a 50 point drop in the dipyridamole group relative to the placebo group

7. Secondary Outcome: Individual Component of Composite Endpoint- Cumulative Ordinal Score
Description: Cumulative sum of WHO Ordinal Scale for Clinical Improvement scores during hospitalization or through 14 days after study drug administration, whichever occurs first. The WHO Ordinal Scale ranges from 1 (no limitation of activities) through 8 (death). By definition, hospitalized patients score 3 or higher on the scale. The equation can be written: Cumulative Ordinal Score = (days in hospital up to 14) x (average ordinal score during hospitalization). Higher scores represent a combination of worse outcomes and longer hospitalizations.
Time Frame: Hospitalization up to 14 days after study drug administration
Population: excluded patients that died or withdrew from the study
Measure: Median (Inter-Quartile Range); unit: score on a scale * days
Arm/Group | Dipyridamole 100 Milligram(mg) | Placebo
Number analyzed (Participants) | 44 | 48
score on a scale * days | 14.3 [9.4 to 21.4] | 15.0 [7.8 to 30.0]
Statistical Analysis 1: Comparison: Dipyridamole 100 Milligram(mg) vs Placebo; Test type: Superiority; p = .95, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: The collection period for adverse events began after informed consent and ended 30 days after administration of the last dose of study drug.
Arm/Group | Dipyridamole 100 Milligram(mg) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/49 | 3/50
Serious Adverse Events (participants affected / at risk) | 14/49 | 30/50
Other Adverse Events (participants affected / at risk) | 43/49 | 15/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dipyridamole 100 Milligram(mg) (N=49) | Placebo (N=50)
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 | 14
Hypotension (Vascular disorders) | 1 | 2
Heart failure (Cardiac disorders) | 1 | 0
Lung infection (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 1
Cardiac Arrest (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Paroxysmal artrial tachycardia (Cardiac disorders) | 0 | 1
Pneumothorax (Musculoskeletal and connective tissue disorders) | 0 | 1
Stroke (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dipyridamole 100 Milligram(mg) (N=49) | Placebo (N=50)
Headache (Nervous system disorders) | 17 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Delirium (General disorders) | 2 | 1
Abdominal pain (General disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 2 | 0
Epistaxis (Vascular disorders) | 2 | 0
Paresthesia (Nervous system disorders) | 1 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Heart failure (Cardiac disorders) | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Edema limbs (Renal and urinary disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Kidney infection (Renal and urinary disorders) | 1 | 0
Atypical urothelial cells in urine (Renal and urinary disorders) | 1 | 0
Incontinence (Renal and urinary disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Emesis (Gastrointestinal disorders) | 1 | 0
Aspartate aminotransferase increased (Gastrointestinal disorders) | 0 | 1
Vaginal hemorrhage (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Ankle pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Body pain (General disorders) | 0 | 1
Fall (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Diaphoresis (General disorders) | 1 | 0
Tremor (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-07-12): https://cdn.clinicaltrials.gov/large-docs/79/NCT04391179/Prot_002.pdf
  • Statistical Analysis Plan (2022-02-03): https://cdn.clinicaltrials.gov/large-docs/79/NCT04391179/SAP_003.pdf